CLINICAL TRIAL: NCT06453954
Title: Evaluating the Effectiveness of the Saving Babies Lives Care Bundle Version 2 on Reducing Perinatal Mortality
Brief Title: Evaluating the Saving Babies Lives Care Bundle Version 2
Acronym: eVOLVE
Status: Completed | Type: Observational
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Dr Alexander Heazell, Professor of Obstetrics, University of Manchester
Other Study IDs: 325846
Record Dates: First submitted 2024-05-21; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Pregnancy Related; Delivery of Health Care
Keywords: Saving Babies Lives Care Bundle Version 2; NHS Maternity Care; Pregnancy; Stillbirth; Perinatal death
MeSH Terms: conditions — Stillbirth; Perinatal Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to learn about the implementation of NHS England's Saving Babies Lives Care Bundle Version 2 to reduce perinatal mortality.

It will explore whether the care bundle is effective at reducing stillbirth rates, neonatal death rates and preterm births in England. It will also explore the lived experiences of women's maternity care and their babies neonatal care, and the views and experiences of healthcare professionals who are involved in delivering the care bundle.

The main questions it aims to answer are:

* Does the care bundle reduce perinatal mortality rates?
* What are women's views and experiences of their maternity and neonatal care?
* What are the barriers around delivering the care bundle and how can this be improved?
* How do health inequalities affect the care women receive?
* How does the workforce culture affect how healthcare professionals use the care bundle?

Perinatal mortality rates and other pregnancy outcomes will be obtained from national data sources. Women and healthcare professionals will be asked to complete a survey and we will interview select groups of participants to further explore their experiences.

Mortality rates will be compared before and after the implementationof the care bundle where data allows. Data from the surveys will be descriptive. Data from the interviews will be analysed using thematic analysis to determine patterns and recurring ideas in the data.

DETAILED DESCRIPTION:
In April 2022, NHS England commissioned the University of Manchester to conduct an independent evaluation of the effectiveness of the Saving Babies' Lives Care Bundle Version 2 (SBLCBv2) on reducing perinatal mortality in England. The study was commissioned in two phases.

Phase 1 comprises a national (service) evaluation of the impact of the SBLCBv2 on perinatal mortality rates, associated clinical outcomes, and any unintended consequences using routine data derived from national databases. Phase 2 comprises a qualitative evaluation to further understand the impact on maternity services, women and their families.

Phase 2 will be conducted in a cohort of maternity units across England using a mixed-methods approach. The views and experiences of women and healthcare professionals towards maternity care in relation to the SBLCBv2 will be sought using surveys and interviews. Additionally, this study will interview organisational leads to assess how resources, leadership and governance may affect implementation in diverse hospital settings.

ELIGIBILITY:
Phase 1:

All births in England.

Phase 2:

Inclusion Criteria:

* women who have given birth in the last 12 months
* women who can understand English
* healthcare professionals involved in delivering the care bundle

Exclusion Criteria:

* women who gave birth more than 12 months ago
* women who cannot understand English
* women without access to the internet for online survey completion
* healthcare professionals not involved in delivering the care bundle

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Phase 1: births in England.
  Phase 2: women who received their antenatal care, labour and birth in 28 participating NHS maternity Trusts in England. Healthcare professionals currently employed in these 28 Trusts.
Sampling Method: Probability Sample
Enrollment: 1773 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Number of stillbirths in England | Up to 60 months
  A baby born after 24 or more weeks completed gestation and which did not, at any time, breathe or show signs of life

SECONDARY OUTCOMES:
Number of babies born preterm | Up to 60 months
  A baby born before 37 weeks gestation
Number of neonatal deaths in England | Up to 60 months
  A live born baby (born at 20+0 weeks gestational age or later, or with a birthweight of 400g or more where an accurate estimate of gestation is not available), who died before 28 completed days after birth
Number of babies born small for gestational age (SGA) | Up to 60 months
  Birthweight less than the 10th percentile for gestational age
Number of women who had a caesarean section | Up to 60 months
  Women delivering by emergency or elective caesarean section
Number of women who had induction of labour | Up to 60 months
  Induced delivieries
Number of women who had an instrumental delivery | Up to 60 months
  Women who had a forceps or ventouse delivery
Number of women who had a spontaneous delivery | Up to 60 months
  Spontaneous delivery without forceps or ventouse delivery
Number of babies admitted to neonatal care | Up to 84 months
  A baby first admitted at the given quarter to any neonatal care unit
Number of babies admitted to neonatal care by gestation | Up to 84 months
  A baby first admitted at the given quarter to a neonatal care unit by gestation weeks at birth
Number of babies admitted to neonatal care by cause of death | Up to 84 months
  A baby first admitted at the given quarter to a neonatal care unit by clinical diagnosis
Number of babies who died whilst on neonatal care | Up to 84 months
  A baby first admitted at any given quarter to a neonatal care unit that died at any point

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Heazell, Prof, Principal Investigator — The University of Manchester
Locations (1):
- Manchester Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
If requested, site-specific data from the questionnaires may be shared with participating NHS Trusts. This data will be provided in an anonymous aggregated format, with only that specific site identified. No identifiable data will be shared with participating NHS Trusts (i.e. names and email addresses will not be shared with NHS sites).
  Following completion of the study, with consent a fully anonymised aggregated dataset [e.g. including anonymous aggregated questionnaire responses] will be deposited in Figshare at the University of Manchester library, which is an open data repository where it will be permanently stored. Researchers at other institutions and others can access the anonymised data directly from the repository and use it for further research or to check our analysis and results. Individual NHS Trusts will not be identified.